CLINICAL TRIAL: NCT01371721
Title: A 6 Month, Open Label, Multi Center, Flexible Dose Extension Study To The B2061014 Study To Evaluate The Safety, Tolerability And Efficacy Of Desvenlafaxine Succinate Sustained Release (Dvs Sr) Tablets In The Treatment Of Children And Adolescent Outpatients With Major Depressive Disorder
Brief Title: A 6-Month Open-Label Extension Study to the B2061014 Study to Evaluate the Safety, Tolerability and Efficacy of DVS SR in the Treatment of Children and Adolescents With MDD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B2061031; 3151A6-3357 (Other: Alias Study Number); 2008-002064-34 (EudraCT Number)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desvenlafaxine Succinate Sustained-Release (Experimental)
  Interventions: Drug: DVS SR

INTERVENTIONS:
Drug: DVS SR — Subjects will receive a flexible-dose of 20, 25, 35 or 50 mg/day as prescribed by the investigator.

SUMMARY:
This is a 6-month, open-label, flexible-dose study evaluating desvenlafaxine succinate sustained release (DVS SR) in the treatment of child and adolescent outpatients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Completed study B2061014 and who in the investigator's opinion would benefit from long term treatment with DVS SR
* Willingness and ability to comply with scheduled visits, treatment plan and procedures

Exclusion Criteria:

* Subject requires precaution against suicide
* Subject not in a generally healthy condition

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2012-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- United States (33):
  - Harmonex Neuroscience Research, Inc., Dothan, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - University of Arizona Clinical and Translational Science Center (CATS), Tucson, Arizona
  - University of Arizona College of Medicine Dept of Psychiatry, Tucson, Arizona
  - Arkansas Psychiatric Clinic Clinical Research Trials, P.A., Little Rock, Arkansas
  - ATP Clinical Research, Incorporated, Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy Clinical Research Center, National City, California
  - Neuropsychiatric Research Center of Orange County, Orange, California
  - Pacific Clinical Research Medical Group, Orange, California
  - Elite Clinical Trials, Incorporated, Wildomar, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Amedica Research Institute, Incorporated, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Kolin Research Group, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute for Behavioral Medicine, LLC, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Lake Charles Clinical Trials,, Lake Charles, Louisiana
  - Precise Research Centers, Flowood, Mississippi
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Incorporated, Las Vegas, Nevada
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Summit Research Network (Oregon), Incorporated, Portland, Oregon
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Focus & Balance, LLC, San Antonio, Texas
  - Grayline Clinical Drug Trials, Witchita Falls, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Rogers Center for Research and Training, Incorporated, Milwaukee, Wisconsin
- Mexico (2):
  - Hospital Aranda de la Parra, S.A. de C.V., León, Guanajuato
  - CIT-Neuropsique, S.C., Monterrey, Nuevo León

REFERENCES:
- [Derived] Atkinson S, Thurman L, Ramaker S, Buckley G, Jones SR, England R, Wajsbrot D. Safety, Tolerability, and Efficacy of Desvenlafaxine in Children and Adolescents with Major Depressive Disorder: Results from Two Open-Label Extension Trials. CNS Spectr. 2019 Oct;24(5):496-506. doi: 10.1017/S1092852918001128. PMID 30419989
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061031&StudyName=A%206-Month%20Open-Label%20Extension%20Study%20to%20the%20B2061014%20Study%20to%20Evaluate%20the%20Safety%2C%20Tolerability%20and%20Efficacy%20of%20DVS%20SR%20in%20the%20Trea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the 8-week, double-blind treatment phase of Desvenlafaxine Succinate Sustained Release (DVS SR B2061014 NCT01372150) and completed the 1-week transition phase (week 9) of the short-term study were eligible to participate in this study (DVS SR B2061031).
Groups:
- Placebo / DVS SR: Placebo in previous study B2061014/DVS SR flexible dose 20 mg - 50 mg in extension study B2061031
- Fluoxetine / DVS SR: Fluoxetine 20 mg in previous study B2061014 /DVS SR flexible dose 20 mg - 50 mg in extension study B2061031
- Desvenlafaxine Succinate Sustained Release / DVS SR: DVS SR weight based (25 mg, 35 mg, 50 mg) in previous study B2061014/DVS SR flexible dose 20 mg - 50 mg in extension study B2061031
Period: Overall Study
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR
Started | 88 | 89 | 92
Treated | 87 | 89 | 92
Completed | 59 | 65 | 62
Not Completed | 29 | 24 | 30
Not completed — Adverse Event | 5 | 4 | 5
Not completed — Protocol Violation | 6 | 4 | 5
Not completed — Lost to Follow-up | 8 | 2 | 6
Not completed — Withdrawal by Subject | 5 | 7 | 11
Not completed — Other | 2 | 3 | 0
Not completed — Lack of Efficacy | 2 | 4 | 3
Not completed — Randomized but not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population - included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Total
Number analyzed (Participants) | 87 | 89 | 92 | 268
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.5 (2.90) | 12.4 (3.01) | 12.8 (3.14) | 12.6 (3.01)
Gender [Count of Participants; unit: Participants]
  Female | 47 | 39 | 49 | 135
  Male | 40 | 50 | 43 | 133

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline at Week 26 in the Children's Depression Rating Scale, Revised (CDRS-R) Total Score Based on Observed Cases
Description: Clinician-rated interview-based scale (with both child and parent or guardian) to assess 17 distinct symptom areas to derive an index of depression severity. Discrepancies between informants' responses were resolved by using most impaired rating given by valid informant. Rated on a 7-point scale; range from 1 (no impairment) to 7 (indicates greater impairment). Total score calculated as sum of the 17 items (range 1 to 119); higher score indicates greater impairment. Adjusted mean presented.
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: ITT-included all randomized participants who had a baseline (of study B2061031) CDRS-R evaluation (Week 9 of study B2061014) took at least 1 dose of study drug and had at least 1 CDRS-R evaluation after the first dose of study drug in the B2061031 study period.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Combination: Combination of 3 groups from previous study B2061014 who received DVS SR flexible dose 20 mg - 50 mg in extension study B2061031
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 55 | 61 | 56 | 172
Score on a Scale | -5.55 (10.80) | -6.41 (11.50) | -5.32 (7.29) | -5.78 (10.03)

2. Secondary Outcome: Change From Baseline at Week 26 in the Clinical Global Impression of Severity (CGI-S) Score Based on Observed Cases
Description: A 7-point clinician rated scale to assess severity of participant's current illness state; range: 1 (normal - not ill at all) to 7 (among the most extremely ill patients). Higher score = more affected. Change: score at observation minus score at baseline. Adjusted mean presented.
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 55 | 61 | 56 | 172
Score on a Scale | -0.78 (1.23) | -0.77 (1.16) | -0.82 (0.92) | -0.79 (1.10)

3. Secondary Outcome: Percentage of Participants With a Clinical Global Impression, Improvement (CGI-I) Response Defined as a Score of 'Very Much Improved' or 'Much Improved' at Week 26
Description: A 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Higher score = more affected.
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 55 | 61 | 56 | 172
Percentage of Participants | 90.9 | 93.4 | 92.9 | 92.4

4. Secondary Outcome: Percentage of Participants With Remission as Determined by a CDRS-R Score of ≤28 at Week 26 Based on Observed Cases
Description: as for outcome 1
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 55 | 61 | 56 | 172
Percentage of Participants | 74.5 | 78.7 | 73.2 | 75.6

5. Primary Outcome: Percentage of Participants Experiencing a Treatment Emergent Adverse Event
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: Safety Population-includes all treatment-assigned participants who took at least one dose of investigational product in the period of study B2061031.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 87 | 89 | 92 | 268
Percentage of Participants | 70.1 | 75.3 | 73.9 | 73.1

6. Secondary Outcome: Percentage of Participants by Clinical Global Impression Improvement (CGI-I) Score at Week 26 Based on Observed Cases
Description: A 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Higher score = more affected.
Time Frame: Week 9 (B2061014)/Day 1 (B2061031) to Week 26 of the B2061031 Study
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Number analyzed (Participants) | 55 | 61 | 56 | 172
Percentage of Participants
  Very Much Improved | 63.6 | 63.9 | 57.1 | 61.6
  Much Improved | 27.3 | 29.5 | 35.7 | 30.8
  Minimally Improved | 3.6 | 3.3 | 5.4 | 4.1
  No Change | 3.6 | 1.6 | 1.8 | 2.3
  Minimally Worse | 0.0 | 1.6 | 0.0 | 0.6
  Much Worse | 1.8 | 0.0 | 0.0 | 0.6
  Very Much Worse | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) recorded from informed consent and assent through Week 30 and Serious Adverse events (SAEs) collected through Week 32 visit. Participants discontinuing prior to Week 28 visit, AEs collected for 14 days and SAEs for 28 days.
Description: Same event may appear as both an AE and an SAE.Data presented are distinct events.Aneven may be categorized as serious in 1 participant and non-serious in another or 1 participant may have experienced both a serious and non-serious event during study.Safety population included all randomized participants receiving at least 1 dose of study drug
Arm/Group | Placebo / DVS SR | Fluoxetine / DVS SR | Desvenlafaxine Succinate Sustained Release / DVS SR | Combination
Serious Adverse Events (participants affected / at risk) | 5/87 | 2/89 | 3/92 | 10/268
Other Adverse Events (participants affected / at risk) | 47/87 | 61/89 | 62/92 | 170/268
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo / DVS SR (N=87) | Fluoxetine / DVS SR (N=89) | Desvenlafaxine Succinate Sustained Release / DVS SR (N=92) | Combination (N=268)
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 1
Frustration (Psychiatric disorders) | 1 | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Self injurious behaviour (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 3 | 1 | 1 | 5
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo / DVS SR (N=87) | Fluoxetine / DVS SR (N=89) | Desvenlafaxine Succinate Sustained Release / DVS SR (N=92) | Combination (N=268)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3 | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 8 | 7 | 22
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 2 | 10
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 3 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 3 | 4
Nausea (Gastrointestinal disorders) | 9 | 14 | 8 | 31
Vomiting (Gastrointestinal disorders) | 5 | 9 | 6 | 20
Fatigue (General disorders) | 2 | 3 | 3 | 8
Bronchitis (Infections and infestations) | 0 | 1 | 4 | 5
Gastroenteritis (Infections and infestations) | 2 | 3 | 2 | 7
Gastroenteritis viral (Infections and infestations) | 4 | 3 | 5 | 12
Influenza (Infections and infestations) | 5 | 1 | 1 | 7
Nasopharyngitis (Infections and infestations) | 11 | 4 | 6 | 21
Pharyngitis (Infections and infestations) | 1 | 2 | 4 | 7
Pharyngitis streptococcal (Infections and infestations) | 2 | 2 | 3 | 7
Sinusitis (Infections and infestations) | 2 | 3 | 3 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 9 | 8 | 24
Viral infection (Infections and infestations) | 0 | 3 | 1 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 2 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 5
Blood pressure increased (Investigations) | 0 | 3 | 3 | 6
Weight increased (Investigations) | 7 | 11 | 12 | 30
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 1 | 5
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 6
Dizziness (Nervous system disorders) | 5 | 5 | 8 | 18
Headache (Nervous system disorders) | 12 | 16 | 19 | 47
Insomnia (Psychiatric disorders) | 2 | 5 | 0 | 7
Irritability (Psychiatric disorders) | 3 | 3 | 2 | 8
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 4 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1 | 10
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The PI must remove any previously undisclosed Confidential Information (other than the Study results themselves) before public release.